CLINICAL TRIAL: NCT05479279
Title: Effectiveness of Neck Stabilization Training Program in Management of Text Neck Syndrome Among Smart Gadget Users
Brief Title: Effectiveness of Neck Stabilization Training Program With Conventional Therapy in Management of Text Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zainab Noor Qazi
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Neck Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Stabilization Training Program (Experimental): Patient education Tens Hot pack Cervical muscle stretching trigger/ tender point release postural re-education cranio-cervical isometrics training of intrascapular, shoulder and upper extremity musculature resistance training with theraband
  Interventions: Other: Neck Stabilization Training Program
- Conventional physical therapy (Active Comparator): Patient education Tens Hot pack Cervical muscle stretching trigger/ tender point release
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Neck Stabilization Training Program — 3 times a week stretching exercises approximately 10 mins dumb bell exercises - 2 sets of 15 reps with weights varying from 1 to 2 kg cranio-cervical isometrics for 10 sec with 15 sec breaks between holds with 10-15 reps Tens 5-10 mins Hotpack 5-10 mins neck stretches home plan - 5 reps/set, 3 sets/ day
  Arms: Neck Stabilization Training Program
Other: Conventional physical therapy — Tens 5-10 mins Hotpack 5-10 mins neck stretches home plan - 5 reps/set, 3 sets/ day
  Arms: Conventional physical therapy

SUMMARY:
1. To compare the effectiveness of neck stabilization training program with conventional physical therapy in management of neck pain and disability in individuals with text neck syndrome.
2. To compare the effectiveness of neck stabilization training program with conventional physical therapy in improving muscle strength and range of motion of cervical spine in individuals with text neck syndrome.

DETAILED DESCRIPTION:
The text neck syndrome was described as a compilation of signs and symptoms due to the repetitive load, stress and pain in the body regions including; neck, shoulder joints, shoulder muscles, and thoracic region initiated by the excessive usage of smartphones for the prolonged time. The text neck syndrome is also called as 'Turtle neck neck syndrome' or 'anterior head syndrome.

Neck flexion in forward direction for using any smart phone could directly affects the cervical and upper thoracic spine. It is stated that increased tilt of the head forward to fifteen degrees exaggerate about 13 Kgs of mechanical force on the cervical spine.

Likewise it progresses to 18 Kgs at 30 degrees, 23 Kgs at 45 degrees and 28 Kgs at 60 degrees of forward neck flexion. The pathological consequences caused by incase of not managing the text neck could be alike to occupational overuse disease or repetitive stress and strain pathology.

ELIGIBILITY:
Inclusion Criteria:

* Gender (both men and women)
* Age: 18-30 years
* Participants using smart phones, laptops and tablets with screen time >3 hours daily, for >6 months.
* Patient diagnosed with text neck syndrome
* Trigger points in cervical muscles (trapezius, levator scapulae and scalene muscles)

Exclusion Criteria:

* Patient diagnosed with neck pain other than text neck syndrome

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 6th week
  It is a functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The test can be interpreted as a raw score, with a maximum score of 50, or as percentage. Highest the score or percentage, higher will be disability.
NPRS | 6th week
  It is a segmented numeric scale in which respondent selects a whole number (0-10). The best reflects the intensity of pain.
Range of motion | 6th Week
  ROM of cervical flexion, extension, lateral rotation and side bending will be measured by universal goniometer.
Cranio-vertebral angle | 6th Week
  This angle is identified as intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No